CLINICAL TRIAL: NCT03754023
Title: The Potential Role of Biomarkers (Urine TIMP-IGFBP7) in Determining the Incidence of Acute Kidney Injury (AKI) in All-comers Patients Presenting to the Emergency Department With Acute Diseases
Brief Title: Biomarker Rule in/Out in Patients With Acute Diseases for Validation of AKI (BRAVA) Acute Kidney Injury
Acronym: BRAVA
Status: Completed | Type: Observational
Sponsor: GREAT Network Italy (Network)
Responsible Party: Sponsor
Other Study IDs: BRAVA Study
Record Dates: First submitted 2018-11-12; First posted 2018-11-27 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2018-11

CONDITIONS: Acute Kidney Injury
Keywords: AKI; Biomarkers; Urine TIMP-IGFBP7; Emergency Department
MeSH Terms: conditions — Acute Kidney Injury; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Urine-TIMP-IGFBP7 biomarker for AKI — Urine-TIMP-IGFBP7 biomarker for AKI

SUMMARY:
The presence or development of AKI impacts on outcomes in patients presenting with acute conditions to the ED. As a result, treating physicians are often concerned with the risk of AKI and take such risk in consideration when making subsequent therapeutic and diagnostic decisions which may result in delaying or withholding therapeutic measures in order to prevent further kidney damage (i.e. avoid imaging studies with contrast media).

If clinicians could be informed early that a patient is at minimal risk for AKI, they could deploy timely and optimal diagnostic and treatment procedures for the underlying disease of the patient without major concerns for causing or exacerbating kidney damage

DETAILED DESCRIPTION:
In patients with acute diseases, it is mandatory for ED Physicians to immediately detect the presence of AKI or exclude; but unfortunately Serum creatinine (SCr) variations (based on KDIGO or AKIN criteria), take 24 to 48 hours to manifest the presence of acute renal ongoing damage. AKI is currently, infact, defined as an increase in SCr of 1.5-fold from baseline within 24 to 48 hours, and decrease in diuresis from admission in hospitalization, using KDIGO.

As consequence, similarly to other biomarkers, such as troponins in acute coronary syndrome and D-dimer in pulmonary embolism, a laboratory test to rule in or rule out AKI is needed in critical patients in ED and our primary objective would be to evaluate the role of urine TIMP-IGFBP7 in this setting.

Primary Objective of the BRAVA Study would be to evaluate the role of the urine biomarkers TIMP-IGFBP7 in predicting the occurrence of AKI in patients presenting to ED with different acute diseases and need for hospitalization.

ELIGIBILITY:
Patient Inclusion Criteria

* Age ≥ 21 years
* >30% risk of developing AKI based on treating physicians' clinical evaluation AND/OR Presence of ONE OF the following conditions:
* Suspected or confirmed sepsis.
* Acute decompensated heart failure.
* Prolonged gastrointestinal losses from vomiting or diarrhea
* Major trauma
* Major bleeding (e.g. gastrointestinal, pulmonary, genitourinary)
* Severe burns
* Diabetic crisis (DKA, HHS)
* Decompensated liver cirrhosis
* Acute coronary syndrome
* Emergent need for iodinated contrast studies
* Shock from any cause

Patient Exclusion Criteria

* Age < 21 years.
* Unable to give informed consent
* Undergoing hemodialysis or peritoneal dialysis
* Pregnancy
* Terminal illness with < 6 months prognosis
* Do-not-resuscitate status

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED who are determined to be at high risk for AKI.
Sampling Method: Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of urine TIMP-IGFBP7 as early biomarker in ruling in or ruling out acute kidney damage in patients presenting to ED with acute diseases. | 48 hours

SECONDARY OUTCOMES:
Overall length in days of hospital stay | 30 hours
Incidence of chronic kidney disease (CKD) | 30 days
Overall mortality | 30 days
Regional (different countries in Asia Pacific Region) incidence of AKI in a cohort of patients presenting to the ED with acute diseases | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Di Somma, Study Director — GREAT Network Italy
Locations (5):
- Prince of Wales Hospital, Sydney, Australia
- Yashoda Hospital, Hyderabad, India
- National University Hospital, Singapore, Singapore
- Konkuk University Medical Center, Seoul, South Korea
- Rhamathibody Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available

REFERENCES:
- [Background] Ostermann M, Joannidis M. Acute kidney injury 2016: diagnosis and diagnostic workup. Crit Care. 2016 Sep 27;20(1):299. doi: 10.1186/s13054-016-1478-z. PMID 27670788
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Wetz AJ, Richardt EM, Wand S, Kunze N, Schotola H, Quintel M, Brauer A, Moerer O. Quantification of urinary TIMP-2 and IGFBP-7: an adequate diagnostic test to predict acute kidney injury after cardiac surgery? Crit Care. 2015 Jan 6;19(1):3. doi: 10.1186/s13054-014-0717-4. PMID 25560277